CLINICAL TRIAL: NCT01157988
Title: Phase II Study of 90Y-ibritumomab Tiuxetan Treatment as a Consolidation After 6th R-CHOP Chemotherapy in Patients With Limited-stage, Bulky Diffuse Large B Cell Lymphoma
Brief Title: 90Y-ibritumomab Tiuxetan Consolidation After 6th R-CHOP Chemotherapy in Patients With Bulky Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Asan Medical Center (Other); Chonbuk National University Hospital (Other); Dong-A University Hospital (Other); Pusan National University Hospital (Other); Severance Hospital (Other)
Responsible Party: Je-Jung Lee, Chonnam National Hwasun Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISL-2007
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2006-04

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: bulky diffuse large B cell lymphoma; 90Y-ibritumomab tiuxetan; clinical response; Safety and toxicity
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ibritumomab tuixetan, response, toxicity (Experimental)
  Interventions: Drug: ibritumomab tiuxetan (Zevalin)

INTERVENTIONS:
Drug: ibritumomab tiuxetan (Zevalin) — During Zevalin treatment, rituximab 250 mg/m2 will be administered with the same methods mentioned above on days 1 and 8. On day 8, within 4 hours following completion of the rituximab dose, 90Y Zevalin at a dose of 0.4 mCi/kg actual body weight for patients with a platelet count > 150,000/L and 0.3 mCi/kg actual body weight for patients with a platelet count of 100,000 - 149,000/L will be injected intravenously over a period of 10 minutes. The maximum allowable dose of 90Y Zevalin is 32 mCi regardless of the patient's body weight. 90Y Zevalin should be administered within 4 hours after radiolabeling of Zevalin with 90Y.

SUMMARY:
This phase II study is aimed at the clinical efficacy and toxicity of 6th R-CHOP chemotherapy followed by ibritumomab tiuxetan (Zevalin) consolidation in patients with limited-stage, bulky diffuse large B cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
The patients with limited-stage, bulky diffuse large B cell lymphoma (DLBCL) are known to have a poor prognosis as like to those with advanced disease. However, there are very limited studies to compare the clinical outcome of therapy after chemotherapy only with combined modality using radiation. Defining local failure at bulky sites as one component of relapse, radioimmuotherapy appears to reduce the failure rates at previous bulky sites. We assessed the clinical efficacy and toxicity of 6th R-CHOP chemotherapy and followed by ibritumomab tiuxetan (Zevalin) consolidation in patients with limited-stage, bulky DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed CD20+ DLBCL
* Patients with stage I/II
* Bulky disease defined by maximum diameter greater than 10 cm or any mediastinal mass exceeding 1/3 the maximum trans- thoracic diameter (more than 8 cm)
* Patients that achieved a complete (CR) or partial response (PR) after 6th R-CHOP chemotherapy
* Aged over 18 years
* ECOG performance status 0-2.

Exclusion Criteria:

* Previous history of chemotherapy for diffuse large B cell lymphoma
* Prior myeloablative therapy
* Prior external-beam radiation to >25% of active bone marrow
* Pregnancy and lactation
* >25% bone marrow infiltration
* Platelet counts <100 000/µl, neutrophil counts <1500/µl
* Children and adolescents under 18 years of age
* Presence of CNS involvement with diffuse large B cell lymphoma
* Positive HIV serology
* Seriously uncontrolled, current infections or other concomitant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Objective response | Up to 24 weeks after the infustion of 90Y-ibritumomab tiuxetan
  Patients receive six cycles of R-CHOP chemotherapy per 21-day intervals. Patients with clearly documented progressive disease will be taken off the study when progression is noted. Patients who achieved a complete or partial response after 6th R-CHOP chemotherapy will receive ibritumomab tiuxetan treatment as a consolidation.
Safety and toxicity | 3 years after the infusion of 90Y-ibritumomab tiuxetan
  After Zevalin treatment, safety profiles will be evaluated with physical examination, vital signs, performance status, serum chemistry and electrolytes, and lymphocytes subset using NCI Common Terminology Criteria for Adverse Events version 3.0, every 4 weeks for 6 months, and then every 3 months for the next 6 months.

SECONDARY OUTCOMES:
Progression-free survival | the time from start of R-CHOP to the first recording of disease progression or death of any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do, South Korea

REFERENCES:
- [Derived] Yang DH, Kim WS, Kim SJ, Kim JS, Kwak JY, Chung JS, Oh SY, Suh C, Lee JJ. Pilot trial of yttrium-90 ibritumomab tiuxetan consolidation following rituximab, cyclophosphamide, doxorubicin, vincristine and prednisolone chemotherapy in patients with limited-stage, bulky diffuse large B-cell lymphoma. Leuk Lymphoma. 2012 May;53(5):807-11. doi: 10.3109/10428194.2011.635857. Epub 2011 Dec 7. PMID 22035417